CLINICAL TRIAL: NCT01022034
Title: Pexy vs. No Pexy in Abdominal Surgery for Full Thickness Rectal Prolapse in Adults: A Randomized Controlled Trial
Brief Title: Pexy Versus Non-pexy for Full Thickness Rectal Prolapse
Acronym: Bergamaschi
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Responsible Party: Roberto Bergamaschi MD, PhD, FRCS, State Univeristy of New York , Stony Brook
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Berg.2007
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Rectal Prolapse
Keywords: Rectal prolapse; mesh; recurrence
MeSH Terms: conditions — Rectal Prolapse; Recurrence | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Pexy group (Active Comparator): This group of patients with full thickness rectal prolapse will receive standard sacral rectopexy with mesh or sutures
  Interventions: Procedure: sacral rectopexy with sutures or meshes
- Non-pexy group (Sham Comparator): These patients will receive full rectal mobilization from the sacrum but without rectopexy
  Interventions: Procedure: full rectal mobilization from the sacrum without sacral rectopexy

INTERVENTIONS:
Procedure: sacral rectopexy with sutures or meshes
  Arms: Pexy group
Procedure: full rectal mobilization from the sacrum without sacral rectopexy
  Arms: Non-pexy group

SUMMARY:
No randomized controlled trial (RCT) has compared no rectopexy to rectopexy for external full-thickness rectal prolapse (FTRP). This study was performed to test the hypothesis that recurrence rates for FTRP following no rectopexy are not inferior to those for rectopexy.

Method: This is a multicenter randomized non-inferiority trial. Eligible patients were randomized to no rectopexy or rectopexy. The no rectopexy arm was defined as abdominal surgery with rectal mobilization only. The rectopexy arm was defined as abdominal surgery with mobilization and pexy. Sigmoid resection was not randomized and was added in the presence of constipation. The endpoint was recurrence rates defined as presence of external FTRP after surgery. A pre-RCT meta-analysis suggested a sample size of 251 patients based on a 15% expected difference in the 5-year cumulative recurrence rate. Recurrence-free curves will be generated and compared using the Kaplan-Meier method and log-rank test, respectively. A Bonferroni adjustment was used. An adjusted p value of <0.01 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* mental ability to understand the procedure
* age range 18 to 70
* both sex

Exclusion Criteria:

* patients with recurrent rectal prolapse
* previous pelvic or colorectal surgery
* previous operation for fecal incontinence
* Cancer
* chronic intestinal Inflammatory diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2003-01; Primary Completion 2009-01 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
long term recurrence of the rectal prolapse | after 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Stony brook University, New York, New York, United States